CLINICAL TRIAL: NCT01169272
Title: Clinical Evaluation Of SonR Atrial Lead In Paradym RF Device SORIN GROUP'S New ICD Plateform
Brief Title: Clinical Evaluation Of The SonR Atrial Lead In Paradym RF Device
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SonR Study - ITSY05
Record Dates: First submitted 2010-07-20; First posted 2010-07-26 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Heart Failure
Keywords: ICD CRT 9770 - PARADYM RF ICD - SonR atrial lead
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CRT-SonR 9770 (Experimental): Active implantable defibrillator with ability to cardiac resynchronization therapy
  Interventions: Device: CRT-SonR 9770

INTERVENTIONS:
Device: CRT-SonR 9770 — Active implantable defibrillator with capacity of cardiac resynchronization therapy
  Other Names: 9770

SUMMARY:
Sorin Group has developed a new atrial lead which is under evaluation during this study. The SonR atrial lead presents a new sensor in the tip of the lead and allows a new feature; interventricular (VV) and atrioventricular (AV) delay (VVD and AVD) optimization.

The new RV autothreshold algorithm has been implemented in the CRT-ICD and will help the physician in his diagnosis avoiding potential lost of capture.

The ICD device has also the capability to be remotely interrogated through the remote monitoring system whose performances will be reported during the study.

Finally, the study will report the electrical and handling performances of the new left ventricular lead.

DETAILED DESCRIPTION:
In this study, the sponsor aims at:

* Demonstrating the safety of the atrial SonR lead;
* Demonstrating the performances of the right ventricular autothreshold algorithm ;
* Reporting the adverse events documented in the study;
* Reporting electrical performances of Sorin Group PARADYM ICD, in order to validate that the performances of those devices are in conformance with longevity and effectiveness objectives;
* Reporting the Sorin atrial SonR and Situs 2 MV left ventricular leads performances;
* Reporting the SonR atrial lead mechanical handling.
* Reporting all information from SonR sensor to validate the SonR data exploitation and the AVD/VVD optimization.
* Reporting the Situs 2 MV LV lead mechanical handling.
* Assessing the user satisfaction (patient and physician) of the remote monitoring solution and the overall availability of the system in terms of data.

Thus, this study intends to show that PARADYM RF ICD operate safely and appropriately in intended-use as part of an ICD system.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for implantation of a CRT 9770 device accordingly to the relevant currently-approved ACC/AHA/ESC guidelines or any relevant currently approved local guidelines for the implantation or replacement of triple-chamber ICD
* Implanted with atrial SonR lead
* Signed and dated informed consent

Exclusion Criteria:

* VT/VF is associated with drug toxicity, electrolyte imbalance, hypoxia, or other reversible cause;
* VT/VF occurred during the acute phase of infarction (< 3 weeks) or during an unstable ischemic phase;
* VF was caused by electrocution;
* Incessant VT/VF;
* Patient is unable to attend the scheduled follow-ups at the implanting centre;
* Patient is already enrolled in another ongoing clinical study;
* Patient is unable to understand the aim of the study and its procedure;
* Patient refuses to cooperate;
* Patient is unable or refuses to provide informed consent;
* Patient is minor (less than 18-year old);
* Patient is pregnant;
* Patient has life expectancy of less than 1 year;
* Patient is forfeiture of freedom or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the SonR lead safety | 3 months
  Complication free rate of the SonR lead superior to 90 %

SECONDARY OUTCOMES:
Incidence of adverse events | 12 months
  Any adverse will be documented thoughout the study and will be reported.
ICD electrical performances | 12 months
  Report all ICD electrical performances of the Paradym RF ICD
Evaluation of the SonR atrial lead performance | 3 months
  Report electrical performances and lead handling at implant
Evaluation of the AV/VV delays optimization | 3 months
  Describe the performances of the manual and automatic AV/VV optimization algorithms. An optional daily life test could be performed to evaluate the automatic optimization at exercise.
Evaluation of the left ventricular lead performances | 12 months
  Report the electrical performances and lead mechanical handling at implant.
Evaluation of the Remote Monitoring Solution | 12 months
  Ensure the Home Monitor setup procedure and daily life use are user friendly for the patient and the back office is convenient for the physician.
Evaluation of the right ventricular autothreshold performances | 1 month
  Demonstrate that the automatic RV pacing thresholds measures are equivalent to the manual test with an authorized error of 0,25V.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe CL Leclercq, Ryhtmologist, Principal Investigator — CHU Rennes
Locations (1):
- Leclercq, Rennes, France